CLINICAL TRIAL: NCT04895917
Title: A Multi-center Open Label Phase II Study of Daratumumab and Pomalidomide in Previously Treated Patients With AL Amyloidosis.
Brief Title: Daratumumab and Pomalidomide in Previously Treated Patients With AL Amyloidosis
Acronym: DarPAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low patient enrollment rate
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Paolo Milani, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-016-IT
Record Dates: First submitted 2021-05-10; First posted 2021-05-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: AL Amyloidosis
Keywords: AL Amyloidosis; Daratumumab; Pomalidomide; relapsed/refractory AL Amyloidosis
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis | interventions — daratumumab; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pomalidomide and daratumumab (Experimental)
  Interventions: Drug: daratumumab and pomalidomide

INTERVENTIONS:
Drug: daratumumab and pomalidomide — Patient eligible to enter the study will receive 6 cycles of 28 days of subcutaneous Daratumumab (1800 mg SC) and oral pomalidomide 4 mg from day 1 to day 21. During cycle 1 and 2, Daratumumab will be administered weekly at days 1, 8, 15, and 22 then from cycle 3 to 6, Daratumumab will be administered every other week at days 1 and 15.

SUMMARY:
This study aims at establishing a new powerful combination of daratumumab and pomalidomide as rescue treatment for patients with R/R AL amyloidosis.

DETAILED DESCRIPTION:
Despite recent advance in understanding the biology of the amyloidogenic clone and despite the availability of different therapeutic options, there are still patients who fail to respond to fist line therapy and experience relapse after response to first line regimens. The toxicity profile of daratumumab resulted favorable in the setting of advanced AL amyloidosis patients with severe organ damage. Pomalidomide has proven to be effective as a single agent in R/R AL amyloidosis with a better safety profile over lenalidomide because of relevant renal toxicity of the latter drug in presence of nephrotic proteinuria. Daratumumab is a recently released mAb that has shown deep hematological responses in R/R multiple myeloma with a favorable toxicity. Up-to-date clinical data have further demonstrated the high efficacy of combination regimens including an ImiD/Daratumumab combination in R/R multiple myeloma reaching unprecedented results in terms of response rate, progression free survival (PFS) and minimal residual disease (MRD) negativity.

On these bases, the present study aims to explore the doublet Daratumumab/pomalidomide in R/R AL amyloidosis. The goal of the study is to obtain rapid, durable and deep hematological responses with a low toxicity profile. The expectation is to attain a very favorable benefit/risk ratio from this combination as these patients should experience a low rate of treatment discontinuation, hospitalization due AEs and/or disease progression and/or organ failures.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of AL amyloidosis;
2. Patients should have received at least one line(and no more than 3 lines)with an alkylating agent and/or a PIn and dexamethasone and not be in VGPR or CR at the time of inclusion (patients who did not reach VGPR or patients in VGPR or better but with an hematological relapse can be included);
3. Measurable hematologic disease: difference between involved and uninvolved FLC > 20 mg/L with an abnormal k/l ratio;
4. Symptomatic organ involvement (heart, kidney, liver/GI tract, peripheral nervous system);
5. Wash-out period of at least 4 weeks from previous antitumor therapy or any investigational treatment or 5 half-lives from previous antibodies, whichever is longer. Treatment from previous therapy should be in accordance to the local clinical practice in which a 4 weeks period is required for the evaluation of response;
6. Adequate bone marrow function prior to 1st drug intake (C1D1), without transfusion or growth factor support within 5 days prior to 1st drug intake, defined as:

   * Absolute neutrophils ≥ 1000/mm3,
   * Platelets ≥ 50000/mm3,
   * Hemoglobin ≥ 9.0 g/dL,
7. Adequate organ function defined as:

   * Serum SGOT/AST or SGPT/ALT < 3.0 X Upper Limit of the normal range (ULN),
   * Serum total bilirubin level<1.5x ULN, unless for subjects with Gilbert's syndrome where the direct bilirubin should then be ≤2.0 x ULN.
8. Female patients who are postmenopausal for at least 1 year before the screening visit, or are surgically sterile, or if they are of childbearing potential, agree to practice effective methods of contraception from the time of signing the informed consent through 30 days after the last dose of study drug, or agree to completely abstain from intercourse (serum pregnancy test has to be performed for all women of childbearing potential at the beginning of each cycle during the study. In addition, a pregnancy test may be done at any time during the study at the discretion of the investigator if a subject miss a period or has unusual menstrual bleeding);
9. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

1. Presence of non-AL amyloidosis;
2. AL amyloidosis with isolated soft tissue involvement;
3. Bone marrow plasma cells >30% and clinically symptomatic multiple myeloma with lytic bone lesions;
4. NT-proBNP >8500 ng/L and hs-troponin I >100 ng/L (cardiac stage IIIb patients);
5. Repetitive ventricular arrhythmias on 24h Holter ECG despite anti-arrhythmic treatment, except if a pacemaker has been implanted;
6. Chronic atrial fibrillation with uncontrolled heart rate;
7. Supine systolic blood pressure <100 mmHg;
8. Subject is a woman who is pregnant, or breast-feeding, or planning to become pregnant;
9. Subjects with known chronic obstructive pulmonary disease or persistent asthma ;
10. Previous anti-CD38 or pomalidomide therapy;
11. Presence of other active malignancy with the exception of non-melanoma skin cancer, cervical cancer, treated early-stage prostate cancer provided that prostate specific antigen is within normal limit, or any completely resected carcinoma in situ;
12. Subjects with known/underlying medical conditions that, in the investigator's opinion would make the administration of the study drug hazardous (ie: uncontrolled diabetes oruncontrolled coronary artery disease);
13. Subject is:

    * (Known to be) seropositive for human immunodeficiency virus (HIV)
    * seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]).Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti- HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
    * (Known to be) seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Rate of good quality (i.e. CR+VGPR) hematologic response. | 6 months
  To assess the rate of good quality (i.e. CR+VGPR) hematologic response at the completion of 6 cycles of Daratumumab plus pomalidomide in patients with relapsed/refractory AL amyloidosis not in VGPR or better after any previous therapy.

SECONDARY OUTCOMES:
To assess in all patients according to their disease history the overall Hematologic Response Rate (CR, VGPR, LowdFLC partial response and PR) at the completion of 1st and 3rd cycles. | At the end of Cycle 1 and Cycle 3 (each cycle is 28 days)
To assess in all patients the overall Hematologic Response Rate including PR at the completion of 6 cycles. | 6 months
To assess in all patients duration of hematologic response. After treatment discontinuation, follow-up will be made to the patient every 3 months for at least 1 year. | 1 year after treatment discontinuation
To assess in all patients the rate of organ response (i.e. cardiac response: NT-proBNB measurement; renal response: proteinuria measurement) and organ improvement, according to standard criteria (Palladini et al JCO 2012, Palladini et al Blood 2014). | 6 months
To assess in all patients the time from the screening to hematologic and organ response. | 6 months
To assess in all patients the hematologic disease progression free survival (PFS) from screening and 1-year PFS from screening (months). | 1 year
To assess in all patients the overall survival (OS) from screening and 1-year OS from screening (months). | 1 year
To assess in all patients the MRD negativity rate according to next generation flow cytometry. | 6 months
To assess quality of life (QoL) using EQ5D-5L. | 1 year after treatment discontinuation

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Policlinico Universitario "Mater Domini", Catanzaro
  - Foundation IRCCS Policlinico San Matteo, Pavia
  - Università Campus Biomedico, Rome